CLINICAL TRIAL: NCT04662749
Title: Influence of Implant Intruding Angle on Osteotome Sinus Elevation Without Grafting
Brief Title: Influence of Intruding Angle on Non-graft Osteotome Sinus Elevation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital of Stomatology, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Feilong Deng, Director, Head of Implantology, Principal Investigator, Clinical Professor, Hospital of Stomatology, Sun Yat-Sen University
Other Study IDs: KQEC-2020-26
Record Dates: First submitted 2020-11-25; First posted 2020-12-10 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-12

CONDITIONS: Partial-edentulism; Osteotome Sinus Lift
Keywords: osteotome sinus lift; endosinus bone gain; sinus floor configuration; intruding angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- concave group: the group whose level of sinus floor is lower than both of the adjacent teeth
- angle group: the group whose level of sinus floor is lower than one of the adjacent teeth and higher than the other one of the adjacent teeth
- flat group: the group whose level of sinus floor is similar to both of the adjacent teeth

SUMMARY:
The contour of maxillary sinus matters in osteotome sinus elevation. So does the implant intruding angle between the axis of the implant and the tangent line of the sinus floor contour. The investigators have been engaged in studying the relationship between the outcome of bone formation and the intruding angle, which could guide our clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Patients with residual bone height >4mm and osteotome sinus elevation together with simultaneous implant placement without grafting

Exclusion Criteria:

* Smokers or patients with systemic disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who visited Guanghua Hospital of Stomatology, Sun Yat-Sen University from July 2006 to August 2018.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2020-02-16 (Actual); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-03-26 (Estimated)

PRIMARY OUTCOMES:
endosinus bone change | from the time of performing the implanting surgery to the latest recalling period, accessed up to 100 months
  endosinus bone change after osteotome sinus elevation without grafting

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Stomatology, Sun Yat-sen University, Guangzhou, Guangdong, China